CLINICAL TRIAL: NCT03309319
Title: A Pilot Study of Rosiglitazone in the Treatment of GH Secreting Pituitary Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhaoyun Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhaoyun Zhang, professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2016-360
Record Dates: First submitted 2017-10-02; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Pituitary Tumor
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Rosiglitazone

ARMS (1):
- Ros (Experimental): Rosiglitazone：2 times a day, 4mg each time（4mgBid）
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — rosiglitazone is added to the primary treatment

SUMMARY:
Growth hormone secreting pituitary adenomas(GHomas) produce excessive GH, stimulating excessive insulin like growth factor 1(IGF-1) synthesis in the liver, thus causing multiple systemic complications. The life expectancy of patients with untreated GHomas is shortened by ten years. The treatment goal of GHomas is to shrink the tumor volume and normalize GH and IGF-1. Under current treatment, only 50-70% of patients get remission. Rosiglitazone is a widely used oral antidiabetic medicine. The investigator's preliminary data showed that rosiglitazone decreased the synthesis of GH and IGF-1 in rat pituitary tumor cells GH3 and hepatocytes respectively. The investigator plan to investigate the efficacy of rosiglitazone in the treatment of patients with GHomas who have not been alleviated by other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GHomas confirmed by surgery
* Patients who did not get biochemical remission: GH nadir after oral glucose tolerance test（OGTT）>1.0ug/L or IGF-1 exceeds age matched normal range

Exclusion Criteria:

* Patients who were allergic to rosiglitazone
* Patients with liver or kidney dysfunction, respiratory failure
* Patients with heart failure
* Patients with edema
* Patients with severe hyperlipidemia
* Patients with osteoporosis or a history of non traumatic fractures
* Patients with pregnancy and lactation
* Patients who had received radiation therapy within 3 years
* Patients who had participated in other clinical trials within 3 months
* Patients with other neoplastic diseases
* Patients with mental and neurological disorders
* Patients with other conditions which were believed not appropriate to take part in the clinical trial

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-10-16 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth hormone(GH) | 6 months
  the decrease of growth hormone(GH)
insulin like factor 1(IGF-1) | 6 months
  the decrease of insulin like factor 1(IGF-1)
tumor volume | 6 months
  the change of tumor volume

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China